CLINICAL TRIAL: NCT05470400
Title: A Phase 1, Open-Label Clinical Trial to Evaluate Safety, Tolerability, and Immunogenicity of Adjuvanted HIV-1 Fusion Peptide Conjugate Vaccine (VRC-HIVVCP0108-00-VP) Alone or in Prime-Boost Regimens With Adjuvanted HIV-1 Envelope Trimer 4571 (VRC-HIVRGP096-00-VP) and HIV-1 Trimer 6931 (VRC-HIVRGP0106-00-VP) Vaccines in Healthy Adults
Brief Title: A Clinical Trial to Evaluate Safety, Tolerability, and Immunogenicity of Adjuvanted HIV-1 Fusion Peptide Conjugate Vaccine Alone or in Prime-Boost Regimens With Adjuvanted HIV-1 Envelope Trimer 4571 and HIV-1 Trimer 6931 Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 303
Record Dates: First submitted 2022-06-29; First posted 2022-07-22 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: HIV
Keywords: HIV; Vaccine; FP conjugate; Trimer 4571; Trimer 6931; Adjuplex; Dose escalation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation - Group 1 (Experimental): Dose Escalation will evaluate the safety, tolerability, and immunogenicity of single adjuvanted doses of the FP conjugate, Trimer 4571 or Trimer 6931 vaccines, in a dose-escalation design. Each product must be assessed as safe prior to use in Prime Boost Regimen.
  Interventions: Biological: FP conjugate vaccine (25 mcg)
- Dose Escalation - Group 2 (Experimental): Dose Escalation will evaluate the safety, tolerability, and immunogenicity of single adjuvanted doses of the FP conjugate, Trimer 4571 or Trimer 6931 vaccines, in a dose-escalation design. Each product must be assessed as safe prior to use in Prime Boost Regimen.
  Interventions: Biological: FP conjugate vaccine (200 mcg)
- Dose Escalation - Group 3 (Experimental): Dose Escalation will evaluate the safety, tolerability, and immunogenicity of single adjuvanted doses of the FP conjugate, Trimer 4571 or Trimer 6931 vaccines, in a dose-escalation design. Each product must be assessed as safe prior to use in Prime Boost Regimen.
  Interventions: Biological: Trimer 6931 (100 mcg)
- Dose Escalation - Group 4 (Experimental): Dose Escalation will evaluate the safety, tolerability, and immunogenicity of single adjuvanted doses of the FP conjugate, Trimer 4571 or Trimer 6931 vaccines, in a dose-escalation design. Each product must be assessed as safe prior to use in Prime Boost Regimen.
  Interventions: Biological: Trimer 6931 (200 mcg)
- Dose Escalation - Group 5 (Experimental): Dose Escalation will evaluate the safety, tolerability, and immunogenicity of single adjuvanted doses of the FP conjugate, Trimer 4571 or Trimer 6931 vaccines, in a dose-escalation design. Each product must be assessed as safe prior to use in Prime Boost Regimen.
  Interventions: Biological: Trimer 4571 (200 mcg)
- Prime Boost Regimen - Group 6 (Experimental): Prime Boost Regimen will evaluate the safety, tolerability, and immunogenicity of adjuvanted vaccines: FP conjugate prime, Trimer 4571 prime, or an FP plus Trimer 4571 prime, all followed by subsequent doses of Trimer 4571, Trimer 6931 and both Trimers combined.
  Interventions: Biological: Trimer 6931 (100 mcg); Biological: Trimer 6931 (200 mcg); Biological: Trimer 4571 (200 mcg); Biological: Trimer 4571 (100 mcg)
- Prime Boost Regimen - Group 7 (Experimental): Prime Boost Regimen will evaluate the safety, tolerability, and immunogenicity of adjuvanted vaccines: FP conjugate prime, Trimer 4571 prime, or an FP plus Trimer 4571 prime, all followed by subsequent doses of Trimer 4571, Trimer 6931 and both Trimers combined.
  Interventions: Biological: FP conjugate vaccine (200 mcg); Biological: Trimer 6931 (100 mcg); Biological: Trimer 6931 (200 mcg); Biological: Trimer 4571 (200 mcg); Biological: Trimer 4571 (100 mcg)
- Prime Boost Regimen - Group 8 (Experimental): Prime Boost Regimen will evaluate the safety, tolerability, and immunogenicity of adjuvanted vaccines: FP conjugate prime, Trimer 4571 prime, or an FP plus Trimer 4571 prime, all followed by subsequent doses of Trimer 4571, Trimer 6931 and both Trimers combined.
  Interventions: Biological: FP conjugate vaccine (200 mcg); Biological: Trimer 6931 (100 mcg); Biological: Trimer 6931 (200 mcg); Biological: Trimer 4571 (200 mcg); Biological: Trimer 4571 (100 mcg)

INTERVENTIONS:
Biological: FP conjugate vaccine (25 mcg) — FP8v1-rTTHC (FP conjugate vaccine) is an HIV-1 fusion peptide conjugated to recombinant tetanus toxoid heavy chain fragment C (rTTHC) via sulfo-SIAB chemical linker.
  Study vaccines will be admixed with Adjuplex adjuvant and administered intramuscularly (IM) via needle and syringe in two injection sites.
  Other Names: FP8v1-rTTHC
  Arms: Dose Escalation - Group 1
Biological: FP conjugate vaccine (200 mcg) — FP8v1-rTTHC (FP conjugate vaccine) is an HIV-1 fusion peptide conjugated to recombinant tetanus toxoid heavy chain fragment C (rTTHC) via sulfo-SIAB chemical linker.
  Study vaccines will be admixed with Adjuplex adjuvant and administered intramuscularly (IM) via needle and syringe in two injection sites.
  Other Names: FP8v1-rTTHC
  Arms: Dose Escalation - Group 2; Prime Boost Regimen - Group 7; Prime Boost Regimen - Group 8
Biological: Trimer 6931 (100 mcg) — HIV-1 Trimer 6931 (Trimer 6931) is a synthetic soluble HIV-1 envelope product that consists of an HIV-1 envelope (Env) trimer variant, derived from consensus clade C sequence (ConC).
  Study vaccines will be admixed with Adjuplex adjuvant and administered intramuscularly (IM) via needle and syringe in two injection sites.
  Other Names: HIV-1 Trimer 6931
  Arms: Dose Escalation - Group 3; Prime Boost Regimen - Group 6; Prime Boost Regimen - Group 7; Prime Boost Regimen - Group 8
Biological: Trimer 6931 (200 mcg) — HIV-1 Trimer 6931 (Trimer 6931) is a synthetic soluble HIV-1 envelope product that consists of an HIV-1 envelope (Env) trimer variant, derived from consensus clade C sequence (ConC).
  Study vaccines will be admixed with Adjuplex adjuvant and administered intramuscularly (IM) via needle and syringe in two injection sites.
  Other Names: HIV-1 Trimer 6931
  Arms: Dose Escalation - Group 4; Prime Boost Regimen - Group 6; Prime Boost Regimen - Group 7; Prime Boost Regimen - Group 8
Biological: Trimer 4571 (200 mcg) — HIV-1 Trimer 4571 (Trimer 4571) is a synthetic soluble HIV-1 envelope product that consists of an HIV-1 envelope (Env) trimer variant, derived from clade A, strain BG505.
  Study vaccines will be admixed with Adjuplex adjuvant and administered intramuscularly (IM) via needle and syringe in two injection sites.
  Other Names: HIV-1 Trimer 4571
  Arms: Dose Escalation - Group 5; Prime Boost Regimen - Group 6; Prime Boost Regimen - Group 7; Prime Boost Regimen - Group 8
Biological: Trimer 4571 (100 mcg) — HIV-1 Trimer 4571 (Trimer 4571) is a synthetic soluble HIV-1 envelope product that consists of an HIV-1 envelope (Env) trimer variant, derived from clade A, strain BG505.
  Study vaccines will be admixed with Adjuplex adjuvant and administered intramuscularly (IM) via needle and syringe in two injection sites.
  Other Names: HIV-1 Trimer 4571
  Arms: Prime Boost Regimen - Group 6; Prime Boost Regimen - Group 7; Prime Boost Regimen - Group 8

SUMMARY:
This is an open-label, dose-escalation study to examine the safety, tolerability, and immunogenicity of adjuvanted Fusion Peptide Vaccine alone or in prime-boost regimens with adjuvanted Trimer 4571 and Trimer 6931 vaccines in healthy adults. The hypothesis is that the vaccines will be safe, and well tolerated when administered alone, and when co-administered with HIV-1 Trimer 4571, in prime-boost regimens, and will induce detectable immune response.

DETAILED DESCRIPTION:
This study has two parts. Part A will evaluate the safety, tolerability, and immunogenicity of single doses of the FP conjugate, Trimer 4571 and Trimer 6931 vaccines, in a dose-escalation design. Each product must be assessed as safe prior to use in Part B. Trimer 4571 with alum adjuvant has been previously evaluated in humans but will be tested in Part A with Adjuplex. Part B will evaluate the safety, tolerability, and immunogenicity of FP conjugate prime, Trimer 4571 prime, or an FP plus Trimer 4571 prime, all followed by subsequent doses of Trimer 4571, or Trimer 6931, or both alone and then both Trimers combined.

Total study duration is 36 months (includes enrollment, planned safety holds and follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to complete the informed consent process, including an Assessment of Understanding (AoU): volunteer demonstrates understanding of this study, completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly.
2. 18-50 years old, inclusive, on day of enrollment.
3. Agrees to comply with planned study procedures and be available for clinic follow-up through the last clinic visit.
4. Agrees not to enroll in another study of an investigational agent during participation in the trial, including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) investigational agents that may subsequently obtain emergency use authorization (EUA) or undergo licensure by the FDA. If a potential participant is already enrolled in a SARS-CoV-2 clinical trial, prior approvals from the SARS-COV-2 study sponsor and HVTN 303 PSRT are required prior to enrollment in HVTN 303.
5. In good general health without clinically significant medical history.
6. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity.
7. Body Mass Index (BMI) ≤ 40.
8. Assessed as low risk for HIV acquisition.
9. Suitable injection sites in the deltoid muscle of each arm, as assessed by a clinician.
10. White blood cells (WBCs) 2,500-12,000/mm3
11. WBC differential either within institutional normal range or approved by the Investigator of Record (IoR) as "not clinically significant."
12. Platelets = 125,000 - 500,000/mm3
13. Hemoglobin

    * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth
    * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth and transgender males who have been on hormone therapy for more than 6 consecutive months
    * ≥ 12.0 g/dL for transgender females who have been on hormone therapy for more than 6 consecutive months
    * For transgender participants who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth
14. Serum creatinine ≤ 1.1 x upper limit of normal (ULN) based on the institutional normal range.
15. Alanine aminotransferase (ALT) ≤1.25 x ULN based on the institutional normal range.
16. Negative for HIV infection by an (US) Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
17. Negative for anti-Hepatitis C antibodies (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV antibodies are detected.
18. Negative for Hepatitis B surface antigen.
19. Agrees to use effective means of birth control from at least 21 days prior to enrollment through 12 weeks after the last product administration.
20. Negative β-HCG (beta human chorionic gonadotropin) pregnancy test (urine or serum) at screening and prior to each study product administration on the day of study product administration.

Exclusion Criteria:

1. Active duty and reserve US military personnel.
2. Breast-feeding or planning to become pregnant from at least 21 days prior to enrollment through 12 weeks after the last product administration.
3. An investigational HIV vaccine (previous placebo recipients are not excluded).
4. Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses ≤ 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment).
5. Blood products within 60 days prior to enrollment
6. Monoclonal antibodies (mAbs), whether licensed or investigational. Exceptions may be made by the HVTN 303 PSRT on a case-by-case basis
7. Receipt of any of the following:

   * Within 4 weeks prior to enrollment:

     * Any licensed live, attenuated vaccine
     * Any adenoviral-vectored SARS-CoV-2 vaccine with FDA Emergency Use Authorization (EUA), FDA licensure or World Health Organization (WHO) Emergency Use Listing (EUL)
   * Within 2 weeks prior to enrollment:

     * Any licensed killed/subunit/inactivated vaccine
     * Any mRNA based or protein SARS-CoV-2 vaccines with FDA EUA, FDA licensure, or WHO EUL
8. Investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
9. Current allergen immunotherapy with antigen injections, unless on maintenance schedule.
10. Current anti-TB prophylaxis or therapy.
11. Serious adverse reactions to vaccines or vaccine components.
12. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
13. Hypertension that is not well controlled.
14. Asthma is excluded if the participant has ANY of the following:

    * Required either oral or parenteral corticosteroids for an exacerbation two or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or co-existing conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
    * Uses more than one medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than one medication for maintenance therapy daily for greater than two years requires PSRT approval.
15. Autoimmune disease, current or history, including psoriasis.
16. Clinically significant immunodeficiency.
17. AESIs: Volunteers who currently have, or have a history of, any condition that could be considered an AESI for the product(s) administered in this protocol.
18. History of generalized urticaria, angioedema, or anaphylaxis. (Not exclusionary: angioedema or anaphylaxis to a known trigger with at least 5 years since last reaction to demonstrate satisfactory avoidance of trigger.).
19. Diabetes mellitus type 1 or type 2.
20. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
21. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
22. Asplenia or functional asplenia.
23. Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study).
24. Any other chronic or clinically significant condition that in the clinical judgement of the investigator would jeopardize the safety or rights of the study participant, including, but not limited to: clinically significant forms of drug or alcohol abuse, serious psychiatric disorders, or cancer that, in the clinical judgement of the site investigator, has a potential for recurrence (excluding basal cell carcinoma).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Troy Martin, Study Chair — HVTN LOC, Fred Hutch; Michael Keefer, M.D., Study Chair — Univ. of Rochester Med. Ctr., HVTU
Locations (6):
- United States (6):
  - Atlanta - Hope Clinic, Atlanta, Georgia
  - BIDMC Vcrs [32077], Boston, Massachusetts
  - New York Blood Center CRS [31801], New York, New York
  - Columbia P&S CRS [30329], New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS [31467], Rochester, New York
  - University of Pittsburgh CRS [1001], Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0): 25 mcg FP Conjugate Vaccine (FP8v1-rTTHC; VRC-HIVVCP0108-00-VP) + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), intramuscularly at Week 0.
- Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0): 200 mcg FP conjugate vaccine (FP8v1-rTTHC; VRC-HIVVCP0108-00-VP) + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), intramuscularly at Week 0.
- Part A, Group 3: 100 mcg Trimer 6931 at w(0): 100 mcg Trimer 6931 (HIV-1 Trimer 6931 Vaccine; VRC-HIVRGP0106-00-VP) + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), intramuscularly at Week 0.
- Part A, Group 4: 200 mcg Trimer 6931 at w(0): 200 mcg Trimer 6931 (HIV-1 Trimer 6931 Vaccine; VRC-HIVRGP0106-00-VP) + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL), intramuscularly at Week 0.
- Part A Group 5: 200 mcg Trimer 4571 at w(0): 200 mcg Trimer 4571 (HIV-1 Trimer 4571 Vaccine; VRC-HIVRGP096-00-VP) + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), intramuscularly at Week 0.
- Part B, Group 6: 200 mcg Trimer 4571 at w(0): 200 mcg Trimer 4571 + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), intramuscularly at Week 0
- Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4): 200 mcg FP conjugate vaccine + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), at Weeks 0 and 4
- Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4): 200 mcg FP conjugate vaccine + 200 mcg Trimer 4571 + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), at Weeks 0 and 4
Period: Overall Study
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Started | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Completed | 2 | 3 | 3 | 3 | 3 | 9 | 10 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9 | 44
Age, Continuous [Median (Full Range); unit: years] | 26 [22 to 27] | 34 [29 to 36] | 42 [22 to 42] | 24 [21 to 38] | 32 [24 to 37] | 25.5 [19 to 32] | 31 [21 to 41] | 37 [18 to 46] | 28.5 [18 to 46]
Age, Customized [Count of Participants; unit: Participants]
  18 - 20 years | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 5
  21 - 30 years | 3 | 1 | 1 | 2 | 1 | 6 | 4 | 1 | 19
  31 - 40 years | 0 | 2 | 0 | 1 | 2 | 2 | 3 | 4 | 14
  41 - 50 years | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 | 1 | 2 | 3 | 1 | 6 | 6 | 5 | 25
  Female | 1 | 1 | 1 | 0 | 1 | 4 | 3 | 4 | 15
  Transgender Male (Female to Male) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Transgender Female (Male to Female) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Gender Queer | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 0 | 1 | 4 | 3 | 4 | 17
  Male | 1 | 1 | 2 | 3 | 2 | 6 | 7 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 1 | 9
  Not Hispanic or Latino | 3 | 3 | 3 | 2 | 1 | 8 | 7 | 8 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
  White | 3 | 3 | 3 | 2 | 1 | 6 | 8 | 8 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through 7 days after each vaccine dose (7 days after the first dose at Week 0 in all Groups, and 7 days after the second dose at Week 4 in Groups 7 and 8 for participants who received the second dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants
  None | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mild | 2 | 2 | 1 | 3 | 2 | 7 | 5 | 4
  Moderate | 1 | 1 | 2 | 0 | 1 | 3 | 5 | 4
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants
  Erythema/Redness: None | 3 | 3 | 3 | 3 | 2 | 9 | 7 | 7
  Erythema/Redness: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Erythema/Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Erythema/Redness: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 6
  Induration/Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Induration/Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 3 | 3 | 3 | 3 | 2 | 9 | 7 | 5
  Erythema and/or Induration: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Erythema and/or Induration: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise a
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants
  Malaise and/or fatigue: None | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
  Malaise and/or fatigue: Mild | 3 | 2 | 2 | 1 | 1 | 7 | 4 | 1
  Malaise and/or fatigue: Moderate | 0 | 1 | 0 | 0 | 1 | 3 | 5 | 6
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 2 | 1 | 2 | 2 | 0 | 3 | 2 | 2
  Myalgia: Mild | 1 | 1 | 1 | 1 | 2 | 4 | 5 | 2
  Myalgia: Moderate | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 4
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 0 | 0 | 1 | 3 | 0 | 3 | 1 | 1
  Headache: Mild | 3 | 2 | 2 | 0 | 3 | 6 | 8 | 4
  Headache: Moderate | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 2 | 2 | 3 | 3 | 3 | 7 | 7 | 3
  Nausea: Mild | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 2
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 2 | 0 | 3 | 3 | 2 | 7 | 1 | 0
  Chills: Mild | 1 | 3 | 0 | 0 | 1 | 2 | 3 | 2
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 4
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 2 | 1 | 3 | 3 | 1 | 5 | 4 | 2
  Arthralgia: Mild | 1 | 2 | 0 | 0 | 2 | 3 | 5 | 3
  Arthralgia: Moderate | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
  Arthralgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms*: None | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms*: Mild | 3 | 1 | 3 | 1 | 2 | 6 | 2 | 1
  Max. Systemic Symptoms*: Moderate | 0 | 2 | 0 | 0 | 1 | 4 | 6 | 5
  Max. Systemic Symptoms*: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Max. Systemic Symptoms*: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 2 | 2 | 3 | 3 | 2 | 8 | 5 | 2
  Temperature: Mild | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 4
  Temperature: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number (Percentage) of Participants With Local Laboratory Values Recorded as Meeting Grade 1 AE Criteria or Above as Specified in the Division of AIDS Table.
Description: The number (percentage) of participants with local laboratory values recorded as meeting Grade 1 AE criteria or above as specified in the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events for alanine aminotransferase (ALT), creatinine, hemoglobin, lymphocyte count, neutrophil count, platelets, white blood cells (WBC) was summarized by treatment arm for each post vaccination time point.
Time Frame: T1-T5: Screening, Days 0,7,14,28; T6: Screening, Days 0,7,14,84,91,98,168,175,182,252,259; T7: Screening, Days 0,7,14,28,35,42,56,63,70,84,91,98,168,175,252,259; T8: Screening, Days 0,7,14,28,35,42,56,63,70,140,147,154,231,238,252
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants
  ALT (U/L) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 8
  ALT (U/L) -Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALT (U/L) -Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 8 | 9
  ALT (U/L) -Day 28 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  ALT (U/L) -Day 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  ALT (U/L) -Day 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT (U/L) -Day 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4
  ALT (U/L) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALT (U/L) -Day 63: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  ALT (U/L) -Day 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 70: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  ALT (U/L) -Day 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  ALT (U/L) -Day 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  ALT (U/L) -Day 91 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 98: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  ALT (U/L) -Day 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  ALT (U/L) -Day 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 147: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  ALT (U/L) -Day 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 154: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  ALT (U/L) -Day 154 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  ALT (U/L) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  ALT (U/L) -Day 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 182: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  ALT (U/L) -Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 231: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  ALT (U/L) -Day 231 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 238: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  ALT (U/L) -Day 238 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 6
  ALT (U/L) -Day 252 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (U/L) -Day 259: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  ALT (U/L) -Day 259 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 8
  Hemoglobin (g/dL) -Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 8 | 9
  Hemoglobin (g/dL) -Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Hemoglobin (g/dL) -Day 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  Hemoglobin (g/dL) -Day 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4
  Hemoglobin (g/dL) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 63: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  Hemoglobin (g/dL) -Day 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 70: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Hemoglobin (g/dL) -Day 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Hemoglobin (g/dL) -Day 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Hemoglobin (g/dL) -Day 91 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 98: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Hemoglobin (g/dL) -Day 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Hemoglobin (g/dL) -Day 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 147: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Hemoglobin (g/dL) -Day 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 154: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Hemoglobin (g/dL) -Day 154 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Hemoglobin (g/dL) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Hemoglobin (g/dL) -Day 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 182: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Hemoglobin (g/dL) -Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 231: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Hemoglobin (g/dL) -Day 231 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 238: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Hemoglobin (g/dL) -Day 238 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 6
  Hemoglobin (g/dL) -Day 252 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL) -Day 259: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Hemoglobin (g/dL) -Day 259 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
  Creatinine (mg/dL) -Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 8
  Creatinine (mg/dL) -Day 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 14 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 8 | 9
  Creatinine (mg/dL) -Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Creatinine (mg/dL) -Day 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  Creatinine (mg/dL) -Day 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4
  Creatinine (mg/dL) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 63: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  Creatinine (mg/dL) -Day 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 70: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Creatinine (mg/dL) -Day 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Creatinine (mg/dL) -Day 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Creatinine (mg/dL) -Day 91 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 98: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Creatinine (mg/dL) -Day 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Creatinine (mg/dL) -Day 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 147: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Creatinine (mg/dL) -Day 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 154: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Creatinine (mg/dL) -Day 154 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Creatinine (mg/dL) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Creatinine (mg/dL) -Day 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 182: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Creatinine (mg/dL) -Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 231: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Creatinine (mg/dL) -Day 231 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 238: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Creatinine (mg/dL) -Day 238 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) -Day 252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 6
  Creatinine (mg/dL) -Day 252 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine (mg/dL) -Day 259: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Creatinine (mg/dL) -Day 259 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WBC (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 8
  WBC (1000 cells/cubic mm) -Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 8 | 9
  WBC (1000 cells/cubic mm) -Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  WBC (1000 cells/cubic mm) -Day 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  WBC (1000 cells/cubic mm) -Day 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4
  WBC (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 63: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  WBC (1000 cells/cubic mm) -Day 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 70: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  WBC (1000 cells/cubic mm) -Day 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  WBC (1000 cells/cubic mm) -Day 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  WBC (1000 cells/cubic mm) -Day 91 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 98: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  WBC (1000 cells/cubic mm) -Day 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  WBC (1000 cells/cubic mm) -Day 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 147: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  WBC (1000 cells/cubic mm) -Day 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 154: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  WBC (1000 cells/cubic mm) -Day 154 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  WBC (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  WBC (1000 cells/cubic mm) -Day 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 182: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 231: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  WBC (1000 cells/cubic mm) -Day 231 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 238: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  WBC (1000 cells/cubic mm) -Day 238 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 6
  WBC (1000 cells/cubic mm) -Day 252 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC (1000 cells/cubic mm) -Day 259: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  WBC (1000 cells/cubic mm) -Day 259 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 8
  Platelets (1000 cells/cubic mm) -Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 8 | 9
  Platelets (1000 cells/cubic mm) -Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Platelets (1000 cells/cubic mm) -Day 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  Platelets (1000 cells/cubic mm) -Day 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4
  Platelets (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 63: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  Platelets (1000 cells/cubic mm) -Day 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 70: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Platelets (1000 cells/cubic mm) -Day 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Platelets (1000 cells/cubic mm) -Day 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Platelets (1000 cells/cubic mm) -Day 91 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 98: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Platelets (1000 cells/cubic mm) -Day 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Platelets (1000 cells/cubic mm) -Day 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 147: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Platelets (1000 cells/cubic mm) -Day 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 154: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Platelets (1000 cells/cubic mm) -Day 154 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Platelets (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Platelets (1000 cells/cubic mm) -Day 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 182: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 231: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Platelets (1000 cells/cubic mm) -Day 231 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 238: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Platelets (1000 cells/cubic mm) -Day 238 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 6
  Platelets (1000 cells/cubic mm) -Day 252 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets (1000 cells/cubic mm) -Day 259: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Platelets (1000 cells/cubic mm) -Day 259 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 8
  Lymphocytes (1000 cells/cubic mm) -Day 7 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 8 | 9
  Lymphocytes (1000 cells/cubic mm) -Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Lymphocytes (1000 cells/cubic mm) -Day 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  Lymphocytes (1000 cells/cubic mm) -Day 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4
  Lymphocytes (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 63: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  Lymphocytes (1000 cells/cubic mm) -Day 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 70: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Lymphocytes (1000 cells/cubic mm) -Day 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 91 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 98: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Lymphocytes (1000 cells/cubic mm) -Day 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 147: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Lymphocytes (1000 cells/cubic mm) -Day 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 154: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Lymphocytes (1000 cells/cubic mm) -Day 154 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 182: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 231: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Lymphocytes (1000 cells/cubic mm) -Day 231 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 238: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Lymphocytes (1000 cells/cubic mm) -Day 238 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 5
  Lymphocytes (1000 cells/cubic mm) -Day 252 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 259: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Lymphocytes (1000 cells/cubic mm) -Day 259 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Screening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 7: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 8
  Neutrophils (1000 cells/cubic mm) -Day 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 8 | 9
  Neutrophils (1000 cells/cubic mm) -Day 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 35: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7
  Neutrophils (1000 cells/cubic mm) -Day 35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 42: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  Neutrophils (1000 cells/cubic mm) -Day 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4
  Neutrophils (1000 cells/cubic mm) -Day 56 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 63: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  Neutrophils (1000 cells/cubic mm) -Day 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 70: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5
  Neutrophils (1000 cells/cubic mm) -Day 70 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Neutrophils (1000 cells/cubic mm) -Day 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Neutrophils (1000 cells/cubic mm) -Day 91 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 98: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Neutrophils (1000 cells/cubic mm) -Day 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Neutrophils (1000 cells/cubic mm) -Day 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 147: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Neutrophils (1000 cells/cubic mm) -Day 147 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 154: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Neutrophils (1000 cells/cubic mm) -Day 154 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Neutrophils (1000 cells/cubic mm) -Day 168 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 175: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Neutrophils (1000 cells/cubic mm) -Day 175 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 182: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 231: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Neutrophils (1000 cells/cubic mm) -Day 231 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 238: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Neutrophils (1000 cells/cubic mm) -Day 238 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 5
  Neutrophils (1000 cells/cubic mm) -Day 252 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils (1000 cells/cubic mm) -Day 259: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 0
  Neutrophils (1000 cells/cubic mm) -Day 259 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply)
Time Frame: 28 days after each vaccine dose (28 days after the first dose at Week 0 in all Groups, and 28 days after the second dose at Week 4 in Groups 7 and 8 for participants who received the second dose).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants
  Mild | 0 | 2 | 1 | 2 | 1 | 1 | 2 | 3
  Moderate | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 2
  Severe | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1
  Potentially life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No AE reported | 2 | 0 | 0 | 1 | 1 | 6 | 5 | 3

6. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: as for outcome 5
Time Frame: as for outcome 5
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants
  Related | 1 | 0 | 2 | 0 | 2 | 2 | 2 | 4
  Not Related | 0 | 3 | 1 | 2 | 0 | 2 | 3 | 2
  No AE reported | 2 | 0 | 0 | 1 | 1 | 6 | 5 | 3

7. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: as for outcome 5
Time Frame: 12 months after each vaccine dose (12 months after the first dose at Week 0 in all Groups, and 12 months after the second dose at Week 4 in Groups 7 and 8 for participants who received the second dose).
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants Reporting Medically Attended Adverse Events (MAAEs)
Description: as for outcome 5
Time Frame: as for outcome 7
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants | 1 | 2 | 1 | 0 | 1 | 3 | 3 | 4

9. Primary Outcome: Number of Participants Reporting Adverse Events of Special Interest (AESIs)
Description: as for outcome 5
Time Frame: as for outcome 7
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: as for outcome 5
Time Frame: as for outcome 7
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3

11. Primary Outcome: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: as for outcome 5
Time Frame: as for outcome 7
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 10 | 10 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Response Rate of Serum Antibody Binding of FP and Envelope Trimer Antigens as Measured by the MSD Assay 2 Weeks After the Last Vaccination.
Description: Meso Scale Discovery Immunogenicity Assay (MSD) was used to measure the IgG binding antibody responses to fusion protein (FP), Trimer 4571, and Trimer 6931 based on two distinct positivity call methods: Method 1, known for its liberal approach, and Method 2, acknowledged for its conservative nature. Method 1 is using the cutoffs from the lab based on the 80 naïve samples (the 95th percentile). Method 2 is using the cutoffs (mean + 3*SD of AUC to each analyte) based on the 80 naïve samples after filtering out %CV>= 30% plus the baseline values from this study. The readout was the area under the curve (AUC) that were calculated from 8 serial dilutions (8-fold) for each sample. Group 5 and Group 6 were combined in the summary of IgG response rate.
Time Frame: Measured at week 2, 2 weeks after the 1st vaccination, for Groups T5+T6, T7, and T8 and week 6, 2 weeks after the 2nd vaccination for Groups T7 and T8.
Population: Overall Number of Participants Analyzed- includes those with samples collected at week 2 for Groups T5+T6, T7, and T8 and week 6 for Groups T7 and T8, who were HIV-uninfected and received the last vaccination. Number Analyzed- counts participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Part A and B, Groups 5+6: 200 mcg Trimer 4571 at w(0): 200 mcg Trimer 4571 + 20% dose/volume (d/v) Adjuplex, to be administered as 0.8 mL, divided into 2 syringes (0.4 mL each), intramuscularly at Week 0
Arm/Group | Part A and B, Groups 5+6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 12 | 8 | 8
Participants
  Fusion Peptide (W2) Positivity call method 1: number analyzed (Participants) | 12 | 7 | 8
  Fusion Peptide (W2) Positivity call method 1 | 1 | 4 | 3
  Fusion Peptide (W2) Positivity call method 2: number analyzed (Participants) | 12 | 7 | 8
  Fusion Peptide (W2) Positivity call method 2 | 1 | 4 | 2
  Fusion Peptide (W6) Positivity call method 1: number analyzed (Participants) | 0 | 3 | 5
  Fusion Peptide (W6) Positivity call method 1 |  | 3 | 5
  Fusion Peptide (W6) Positivity call method 2: number analyzed (Participants) | 0 | 3 | 5
  Fusion Peptide (W6) Positivity call method 2 |  | 3 | 5
  Trimer 4571 (W2) Positivity call method 1: number analyzed (Participants) | 12 | 7 | 8
  Trimer 4571 (W2) Positivity call method 1 | 0 | 1 | 0
  Trimer 4571 (W2) Positivity call method 2: number analyzed (Participants) | 12 | 7 | 8
  Trimer 4571 (W2) Positivity call method 2 | 0 | 0 | 0
  Trimer 4571 (W6) Positivity call method 1: number analyzed (Participants) | 0 | 3 | 5
  Trimer 4571 (W6) Positivity call method 1 |  | 1 | 5
  Trimer 4571 (W6) Positivity call method 2: number analyzed (Participants) | 0 | 3 | 5
  Trimer 4571 (W6) Positivity call method 2 |  | 0 | 3
  Trimer 6931 (W2) Positivity call method 1: number analyzed (Participants) | 12 | 7 | 8
  Trimer 6931 (W2) Positivity call method 1 | 3 | 1 | 2
  Trimer 6931 (W2) Positivity call method 2: number analyzed (Participants) | 12 | 7 | 8
  Trimer 6931 (W2) Positivity call method 2 | 0 | 1 | 0
  Trimer 6931 (W6) Positivity call method 1: number analyzed (Participants) | 0 | 3 | 5
  Trimer 6931 (W6) Positivity call method 1 |  | 1 | 5
  Trimer 6931 (W6) Positivity call method 2: number analyzed (Participants) | 0 | 3 | 5
  Trimer 6931 (W6) Positivity call method 2 |  | 0 | 2

13. Primary Outcome: Magnitude of Serum Antibody Binding of FP and Envelope Trimer Antigens as Measured by the MSD Assay 2 Weeks After the Last Vaccination.
Description: Meso Scale Discovery Immunogenicity Assay (MSD) was used to measure the IgG binding antibody responses to fusion protein (FP), Trimer 4571, and Trimer 6931 based on two distinct positivity call methods: Method 1, known for its liberal approach, and Method 2, acknowledged for its conservative nature. Method 1 is using the cutoffs from the lab based on the 80 naïve samples (the 95th percentile). Method 2 is using the cutoffs (mean + 3*SD of AUC to each analyte) based on the 80 naïve samples after filtering out %CV>= 30% plus the baseline values from this study. The readout was the area under the curve (AUC) that were calculated from 8 serial dilutions (8-fold) for each sample. The Unit of Measure is expressed as Mean Electrochemiluminescence Signal*1/dilution to reflect the AUC of responses across serial dilutions. Group 5 and Group 6 were combined in the summary of IgG magnitudes.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: Mean ECL Signal*1/dilution
Arm/Group | Part A and B, Groups 5+6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
Number analyzed (Participants) | 12 | 8 | 8
Mean ECL Signal*1/dilution
  Fusion Peptide (W2): number analyzed (Participants) | 12 | 7 | 8
  Fusion Peptide (W2) | 447.40 [276.10 to 663.00] | 1462.00 [596.30 to 2334.50] | 557.30 [380.60 to 1216.80]
  Fusion Peptide (W6): number analyzed (Participants) | 0 | 3 | 5
  Fusion Peptide (W6) |  | 9463.00 [7766.80 to 12143.80] | 8568.50 [5487.00 to 10460.50]
  Trimer 4571 (W2): number analyzed (Participants) | 12 | 7 | 8
  Trimer 4571 (W2) | 124.60 [84.70 to 165.30] | 61.70 [56.60 to 118.60] | 87.80 [68.80 to 138.50]
  Trimer 4571 (W6): number analyzed (Participants) | 0 | 3 | 5
  Trimer 4571 (W6) |  | 236.40 [143.20 to 367.20] | 1192.00 [744.50 to 1945.00]
  Trimer 6931 (W2): number analyzed (Participants) | 12 | 7 | 8
  Trimer 6931 (W2) | 175.60 [107.20 to 218.60] | 106.30 [90.90 to 149.40] | 118.70 [99.40 to 179.50]
  Trimer 6931 (W6): number analyzed (Participants) | 0 | 3 | 5
  Trimer 6931 (W6) |  | 103.00 [87.80 to 192.00] | 572.10 [414.70 to 677.50]

ADVERSE EVENTS:
Time Frame: SAEs, medically attended adverse events (MAAEs), adverse events of special interest (AESIs) and AEs leading to early participant withdrawal or permanent discontinuation were collected throughout the study and for 12 months following any receipt of study product. Other unsolicited AEs were collected for 28 days after any receipt of study vaccination. Reactogenicity events (solicited AEs) were collected through 7 full days after each vaccination.
Arm/Group | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) | Part A Group 5: 200 mcg Trimer 4571 at w(0) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 10/10 | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) (N=3) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) (N=3) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) (N=3) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) (N=3) | Part A Group 5: 200 mcg Trimer 4571 at w(0) (N=3) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) (N=10) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) (N=10) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4) (N=9)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: 25 mcg FP Conjugate Vaccine at w(0) (N=3) | Part A, Group 2: 200 mcg FP Conjugate Vaccine at w(0) (N=3) | Part A, Group 3: 100 mcg Trimer 6931 at w(0) (N=3) | Part A, Group 4: 200 mcg Trimer 6931 at w(0) (N=3) | Part A Group 5: 200 mcg Trimer 4571 at w(0) (N=3) | Part B, Group 6: 200 mcg Trimer 4571 at w(0) (N=10) | Part B, Group 7: 200 mcg FP Conjugate Vaccine at w(0, 4) (N=10) | Part B, Group 8: 200 mcg FP Conjugate Vaccine + 200 mcg Trimer 4571 at w(0, 4) (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Solicited) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 6 (6)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (Solicited) (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 9 (9) | 9 (9)
Fatigue (Solicited) (General disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 10 (10) | 10 (10) | 9 (9)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site erythema (Solicited) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (Solicited) (General disorders) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 10 (10) | 10 (10) | 9 (9)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (Solicited) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Solicited) (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 7 (7)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 6 (6) | 7 (7)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 7 (7) | 8 (8) | 7 (7)
Headache (Solicited) (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 7 (7) | 9 (9) | 8 (8)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT05470400/Prot_000.pdf
  • Statistical Analysis Plan: Immunogenicity (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT05470400/SAP_001.pdf
  • Statistical Analysis Plan: Safety (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT05470400/SAP_002.pdf